CLINICAL TRIAL: NCT06775184
Title: The Effect of Fiberoptic Bronchoscopy Examination on Supraglottic Airway Devices Position in Patients Undergoing Elective Surgery
Brief Title: Fiberoptic Bronchoscopy on Supraglottic Airway Devices Position
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, KMUHIRB-F(I)-20240331, Associate professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-F(I)-20240331
Record Dates: First submitted 2025-01-06; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Supraglottic Airway Devices Position
Keywords: supraglottic device; video laryngeal mask; fiberoptic bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Third-generation SADs (SaCoVLM) (Experimental): The third-generation SADs (i.e. SaCoVLM™) combines video system and laryngeal mask with gastric drain.
  Interventions: Device: a native video image system
- Second-generation SADs (I-gel™) (Active Comparator): The second-generation SADs (i.e. I-gel™) with a gastric drain conduit have designed to reduce the risk of gastric reflux and aspiration.
  Interventions: Device: a native video image system; Device: Fiberoptic bronchoscope

INTERVENTIONS:
Device: a native video image system — The visualization of the glottic structures through the SaCoVLM™ imaging system is graded as follows: Grade1: Visibility of the lateral portion of the right epiglottic fold and part of the laryngeal inlet. Grade 2: Visibility of both epiglottic folds and part of the laryngeal inlet. Grade 3: Visibility of the laryngeal inlet and part of the vocal cords. Grade 4: Visibility of the entire vocal cords.
Device: Fiberoptic bronchoscope — The position of the i-Gel is checked using a fiberoptic endoscope
  Arms: Second-generation SADs (I-gel™)

SUMMARY:
A comparison of SaCo VLMTM video laryngeal mask airway with the I-gel supraglottic airway during airway management in patients undergoing elective surgery.

DETAILED DESCRIPTION:
The position of the supraglottic airway is checked using a fiberoptic endoscope: The bronchoscope is placed at the opening of the laryngeal mask, and assessed using the following grading system: Grade 1: Vocal cords not visible. Grade 2: Vocal cords and anterior epiglottis visible. Grade 3: Vocal cords and posterior epiglottis visible. Grade 4: Only vocal cords visible.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I~III, age 18~65 y/o, BMI 18~30kg/m2, elective surgery, surgery duration < 2 hours, supine position, general anesthesia with laryngeal mask airway insertion

Exclusion Criteria:

* Smoking, betel nuts use, any known anatomical variation or disease of facial or airway structure, anticipated difficult airway, limited mouth opening distance or neck motility, loosening teeth, gastroesophageal reflux history, ongoing upper airway infection or inflammation symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
glottic visualization grades by fiberoptic exam assessment | From anesthesia induction to the end of surgery
  Grade 1: vocal cords were not visualizedGrade 2: vocal cords and anterior epiglottis were visualizedGrade 3: vocal cords and posterior epiglottis were visualized Grade 4: vocal cords only were visualized

SECONDARY OUTCOMES:
Intra-operative effectiveness | From anesthesia induction to the end of surgery
  Secondary outcomes were evaluated by oropharyngeal sealing pressure, first attempt success rate, insertion time

IPD SHARING:
Plan to Share IPD: Undecided
not decided